CLINICAL TRIAL: NCT05776966
Title: Increasing Women's Engagement in Medication Treatment for Opioid Use Disorder Through Digital Intervention
Brief Title: Women's Opioid Treatment Follow-up Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Dawn E. Sugarman, PhD, Research Psychologist, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023P000495; K23DA050780 (NIH)
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gender-specific digital intervention plus treatment as usual (GSDI+TAU) (Experimental): GSDI + TAU includes the addition of a gender-specific digital intervention (GSDI) to treatment as usual. The GSDI has a web-based component and a mobile component. The web-based portion of the GSDI includes: (1) gender-specific psychoeducation on substance use disorders, (2) specific education on opioid use disorder, including information about medication treatment for opioid use disorder, and (3) information on relapse-prevention skills. Participants complete the web-based portion immediately after completing baseline assessments. The mobile component includes three parts: (1) weekly self-report surveys of opioid and other substance use and medication adherence, (2) weekly skills-practice exercises, and (3) daily motivational messages encouraging self-care. Participants engage with the mobile component after completing the web-based portion until the end of the study (12 weeks).
  Interventions: Behavioral: Gender-specific digital intervention (GSDI); Other: Treatment as usual
- Treatment as usual (TAU) (Other): TAU for opioid use disorder consists of a mix of medication treatment and individual and group therapy services across various levels of care: inpatient, residential, and outpatient. Residential treatment is for adults who have completed detoxification and require additional treatment in a structured environment. Inpatient treatment includes short-term care and detoxification treatment and incorporates a combination of group, family, and individual therapy targeted at medical stabilization, reducing the severity of the patient's symptoms, and providing resources and ongoing support to prevent relapse. Outpatient treatment is focused on comprehensive evaluation and stabilization.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Gender-specific digital intervention (GSDI) — The GSDI is a digital intervention that incorporates factors that are more prevalent in women with opioid use disorder that may affect their treatment outcomes. The content for the intervention was derived from research on gender-specific substance use disorder antecedents, consequences, and treatment outcomes.
  Arms: Gender-specific digital intervention plus treatment as usual (GSDI+TAU)
Other: Treatment as usual — Participants will receive treatment as usual for opioid use disorder which is a mix of medication treatment and individual and group therapy services across various levels of care.

SUMMARY:
The goal of this study is to examine the feasibility of a gender-specific digital intervention for women with opioid use disorder. In this study, women with opioid use disorder will be randomized to receive treatment-as-usual plus a gender-specific digital intervention or treatment-as-usual only. Feasibility, satisfaction, and engagement with the intervention are the primary outcomes and will be measured post-intervention and at two-week, 6-week, and 12-week follow-up visits.

DETAILED DESCRIPTION:
This study has two aims: (1) to demonstrate the feasibility of delivering a gender-specific digital intervention (GSDI) to women with opioid use disorder; (2) to collect preliminary estimates on the effect of the GSDI on engagement in medication treatment for opioid use disorder (MOUD). The investigators will conduct a pilot randomized controlled trial to achieve these aims. Women (N=40) who have recently initiated MOUD (within 30 days) will be enrolled and randomized to receive either the GSDI+TAU (gender-specific digital intervention + treatment as usual) or TAU-only. Feasibility, satisfaction, and engagement with the GSDI are the primary outcomes and will be measured post-intervention and at two-week, 6-week, and 12-week follow-ups. MOUD engagement will be assessed at two time-points: (1) 6-weeks and (2) 12-weeks post-enrollment to collect preliminary estimates on the effect of the GSDI on MOUD engagement.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years of age or older
* current opioid use disorder diagnosis
* have a smartphone
* initiated medication treatment for opioid use disorder in the past 30 days,
* able to provide informed consent

Exclusion Criteria:

* an acute psychiatric or medical condition, or cognitive impairment, that would impair the ability to complete study procedures
* admitted to their current treatment episode on an involuntary status

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Due to the gender-specific focus of this study, only participants who do identify as women will be included.
Enrollment: 39 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2025-10-16 (Actual); Study Completion 2025-10-16 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | Immediately after the web-based portion of the intervention, Week 12
  The Client Satisfaction Questionnaire (CSQ) assesses participant satisfaction of the digital intervention. The original CSQ has 8 items and we have added an additional 8 items to gather satisfaction with specific aspects of the digital intervention.
System Usability Scale | 12 weeks
  The System Usability Scale (SUS) is a 10-item questionnaire with five response options for respondents from Strongly agree to Strongly disagree. The SUS is used to measure usability of products and services, including hardware, software, mobile devices, websites, and applications.
Engagement metrics | Week 1 - Week 12
  Engagement data will be retrieved from MetricWire including number of logins, number of completed check-ins and skills practices, and time spent on each of these activities. Time spent on the web-based portion of the GSDI will be calculated from REDCap.
Qualitative Exit Interview | Week 12
  Qualitative user experience exit interviews will be coded and analyzed using thematic analysis methodology to identify common themes.

SECONDARY OUTCOMES:
Timeline Followback | Week 2, Week 6, Week 12
  The Timeline Followback calendar method will be used to collect self-report data on medication for opioid use disorder adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No